CLINICAL TRIAL: NCT04777994
Title: A Phase 1 Study With ABBV-CLS-484 Alone and in Combination in Subjects With Locally Advanced or Metastatic Tumors
Brief Title: Study With ABBV-CLS-484 in Participants With Locally Advanced or Metastatic Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-431; 2023-507568-38-00 (Other: EU CT)
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor Cancer
Keywords: Cancer; Tumor; anti-PD-1; ABBV-CLS-484; clear cell renal cell carcinoma (ccRCC); head and neck squamous cell carcinoma (HNSCC); non-small cell lung cancer (NSCLC); relapsed or refractory (R/R); Microsatellite instability - high tumors (MSI-H); Vascular Endothelial Growth Factor Receptor (VEGFR) Tyrosine Kinase Inhibitor (TKI)
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — osunprotafib; Receptors, Vascular Endothelial Growth Factor; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Monotherapy Dose Escalation (Experimental): ABBV-CLS-484 will be administered as a monotherapy in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-484
- Combination Dose Escalation with PD-1 Inhibitor (Experimental): ABBV-CLS-484 will be administered in combination with Programmed Cell Death-1 Inhibitor in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-484; Drug: Programmed Cell Death-1 (PD-1) Inhibitor
- Monotherapy Expansion (Experimental): ABBV-CLS-484 will be administered at the determined recommended dose in subjects with locally advanced or metastatic, relapsed or refractory head and neck squamous cell carcinoma (HNSCC), relapsed or refractory non-small cell lung cancer (NSCLC), and advanced clear cell renal cell carcinoma (ccRCC)
  Interventions: Drug: ABBV-CLS-484
- Combination Expansion with PD-1 Inhibitor (Experimental): ABBV-CLS-484 will be administered at the determined recommended dose in combination with Programmed Cell Death-1 Inhibitor in subjects with locally advanced or metastatic, HNSCC, NSCLC, MSI-H tumors refractory to PD-1/PD-L1, and advanced ccRCC.
  Interventions: Drug: ABBV-CLS-484; Drug: Vascular Endothelial Growth Factor Receptor (VEGFR) Tyrosine Kinase Inhibitor (TKI)
- Combination Dose Escalation with VEGFR TKI (Experimental): ABBV-CLS-484 will be administered in combination with a Vascular Endothelial Growth Factor Receptor (VEGFR) Tyrosine Kinase Inhibitor (TKI) in subjects with solid tumors
  Interventions: Drug: ABBV-CLS-484; Drug: Programmed Cell Death-1 (PD-1) Inhibitor
- Combination Expansion (Experimental): ABBV-CLS-484 will be administered at the determined recommended dose in combination with VEGFR TKI in subjects with locally advanced or metastatic, HNSCC, NSCLC, MSI-H tumors refractory to PD-1/PD-L1, and advanced ccRCC.
  Interventions: Drug: ABBV-CLS-484; Drug: Vascular Endothelial Growth Factor Receptor (VEGFR) Tyrosine Kinase Inhibitor (TKI)

INTERVENTIONS:
Drug: ABBV-CLS-484 — Oral Capsule
Drug: Vascular Endothelial Growth Factor Receptor (VEGFR) Tyrosine Kinase Inhibitor (TKI) — Oral Tablet
  Arms: Combination Expansion; Combination Expansion with PD-1 Inhibitor
Drug: Programmed Cell Death-1 (PD-1) Inhibitor — Intravenous (IV) infusion
  Arms: Combination Dose Escalation with PD-1 Inhibitor; Combination Dose Escalation with VEGFR TKI

SUMMARY:
The study will assess the safety, PK, PD, and preliminary efficacy of ABBVCLS-484 as monotherapy and in combination with a PD-1 targeting agent or with a or a vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor (TKI).

The trial aims to establish a safe, tolerable, and efficacious dose of ABBVCLS-484 as monotherapy and in combination. The study will be conducted in three parts. Part 1 Monotherapy Dose Escalation, Part 2 Combination Dose Escalation and Part 3 Dose Expansion (Monotherapy and Combination therapy).

Part 1, ABBV-CLS-484 will be administered alone in escalating dose levels to eligible subjects who have advanced solid tumors.

Part 2, ABBV-CLS-484 will be administered at escalating dose levels in combination with a PD-1 targeting agent or with a VEGFR TKI to eligible subjects who have advanced solid tumors.

Part 3, ABBV-CLS-484 will be administered alone as a monotherapy at the determined recommended dose in subjects with locally advanced or metastatic, relapsed or refractory head and neck squamous cell carcinoma (HNSCC), relapsed or refractory non-small cell lung cancer (NSCLC), and advanced clear cell renal cell carcinoma (ccRCC). ABBV-CLS-484 will also be administered at the determined recommended dose in combination with a PD-1 targeting or with a VEGFR TKI agent in subjects with locally advanced or metastatic, HNSCC, NSCLC, MSI-H tumors refractory to PD-1/PD-L1, and advanced ccRCC.

ELIGIBILITY:
Inclusion Criteria:

* Must weigh at least 35 kilograms (kg).
* An Eastern Cooperative Oncology Group (ECOG) performance status <= 2.
* Life expectancy of >= 12 weeks.
* Laboratory values meeting protocol criteria.
* QT interval corrected for heart rate < 470 msec (using Fridericia's correction), and no clinically significant electrocardiographic findings.
* Measurable disease defined by RECIST 1.1 criteria.

For Monotherapy and Combination Dose Escalation:

* Participants with histologically or cytologically proven metastatic or locally advanced tumors, for which no effective standard therapy exists, or where standard therapy has failed. Participants must have received at least 1 prior systemic anticancer therapy for the indication being considered.

For Monotherapy Dose Expansion only:

* Participants must have received at least 1 prior line containing PD-1/PD-L1 targeted therapy with a best response by RECIST v1.1 of CR/PR/stable (any duration) or stable disease (for greater than 6 months); AND
* Must have been previously treated with 1 or more prior lines of therapy in the locally advanced or metastatic setting with the following tumor types:

  * Relapsed/refractory HNSCC
  * Relapsed/refractory NSCLC
  * Advanced ccRCC

For PD-1 Targeting Agent Combination Dose Expansion only:

* For the following tumor types, subject must have received at least 1 prior line containing PD-1/PD-L1 targeted therapy with response by RECIST v1.1 of CR/PR (any duration) or stable disease (for greater than 6 months):

  * Relapsed HNSCC
  * Relapsed NSCLC
  * Relapsed Advanced ccRCC
* For the following tumor types, subject must have received at least 1 prior line containing PD-1/PD-L1 targeted therapy and have had disease progression with PD-1/PD-L1 targeted therapy:

  * Locally Advanced or metastatic MSI-H tumors

For VEGFR TKI Combination Dose Expansion only:

* Relapsed advance ccRCC with no more than 1 prior VEGFR TKI
* Participants no recent history of hemorrhage, including hemoptysis, hematemesis, or melena
* Participants with poorly controlled hypertension are excluded.

Exclusion Criteria:

* Untreated brain or meningeal metastases (i.e., subjects with history of metastases are eligible provided they do not require ongoing steroid treatment and have shown clinical and radiographic stability for at least 28 days after definitive therapy)
* Unresolved Grade 2 or higher toxicities related to previous anticancer therapy except alopecia.
* Unresolved Grade 2 or higher peripheral neuropathy.
* History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
* Recent history (within 6 months) of congestive heart failure (defined as New York Heart Association, Class 2 or higher), ischemic cardiovascular event, pericarditis, or clinically significant pericardial effusion or arrythmia.
* Recent history (within 6 months) of Childs-Pugh B or C classification of liver disease.
* History of clinically significant medical and/or psychiatric conditions or any other reason that, in the opinion of the investigator, would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive study drug.
* History of uncontrolled, clinically significant endocrinopathy.
* Known gastrointestinal disorders making absorption of oral medications problematic; subject must be able to swallow capsules.
* If treated with a PD-1/aPD-L1 targeting or other immune-oncology agents in the past, excluded if had prior pneumonitis, prior Grade 3 or higher immune mediated toxicity, hypersensitivity to administered drug or drug related toxicity requiring discontinuation.
* Active autoimmune disease requiring systemic treatment in past 2-years (exceptions for endocrinopathies, vitiligo or atopic conditions).
* History of solid organ transplant or allogeneic stem cell transplant.
* History of other malignancy, with the following exceptions:

  * No known active disease present within >= 3 years before first dose of study treatment and felt to be at low recurrence by investigator.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* History of interstitial lung disease or pneumonitis.
* Major surgery <= 28 days prior to first dose of study drug
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection per local testing practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Maximum Observed Plasma/Serum Concentration (Cmax) Of ABBV-CLS-484 (Monotherapy) | Baseline Up to Approximately Day 42
  Maximum plasma/serum concentration of ABBV-CLS-484
Dose Escalation: Maximum Observed Plasma/Serum Concentration (Cmax) Of Programmed Cell Death-1 (PD-1) Inhibitor (Combination therapy) | Baseline Up to Approximately Day 64
  Maximum plasma/serum concentration of PD-1 inhibitor
Dose Escalation: Maximum Observed Plasma/Serum Concentration (Cmax) Of VEGFRTKI (Combination therapy) Maximum plasma/serum concentration of PD-1 inhibitor | Baseline Up to Approximately Day 64
  Maximum plasma/serum concentration of PD-1 inhibitor
Dose Escalation: Time To Cmax (Tmax) Of ABBV-CLS-484 (Monotherapy) | Baseline Up to Approximately Day 42
  The amount of time taken to reach Cmax
Dose Escalation: Time To Cmax (Tmax) Of PD-1 Inhibitor (Combination therapy) | Baseline Up to Approximately Day 64
  The amount of time taken to reach Cmax
Dose Escalation Time to Cmax (Tmax) of VEGFR TKI (Combination therapy) | Baseline Up to Approximately Day 64
  The amount of time taken to reach Cmax
Dose Escalation: Phase Elimination Rate Half-Life (t1/2) Of ABBV-CLS-484 (Monotherapy) | Baseline Up to Approximately Day 42
  Terminal phase elimination half-life (t1/2)
Dose Escalation: Phase Elimination Rate Half-Life (t1/2) Of PD-1 Inhibitor (Combination therapy) | Baseline Up to Approximately Day 64
  Terminal phase elimination half-life (t1/2)
Dose Escalation: Phase Elimination Rate Half-Life (t1/2) Of VEGFR TKI (Combination therapy) | Baseline Up to Approximately Day 64
  Terminal phase elimination half-life (t1/2)
Dose Escalation: Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of ABBV-CLS-484 (Monotherapy) | Baseline Up to Approximately Day 42
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Dose Escalation: Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of PD-1 Inhibitor (Combination therapy) | Baseline Up to Approximately Day 64
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Dose Escalation: Area Under The Plasma Or Serum Concentration-Time Curve (AUC) Of VEGFR TKI (Combination therapy) | Baseline Up to Approximately Day 64
  AUC is the area under the serum concentration versus time curve of the last measurable concentration prior to next dose
Dose Escalation: Recommended Phase 2 Dose (RP2D) and/or Maximum Tolerated Dose of ABBV-CLS-484 | Baseline Up to Approximately Day 42
  The MTD and/or RP2D of ABBV-CLS-484 will be determined during the monotherapy therapy dose escalation phase of the study
Dose Escalation: Recommended Phase 2 Dose (RP2D) and/or Maximum Tolerated Dose of ABBV-CLS-484 and a PD-1 Inhibitor (Combination therapy) | Baseline Up to Approximately Day 64
  The MTD and/or RP2D of ABBV-CLS-484 and PD-1 inhibitor will be determined during the combination therapy dose escalation phase of the study
Dose Escalation: Recommended Phase 2 Dose (RP2D) and/or Maximum Tolerated Dose of ABBV-CLS-484 and a VEGFR TKI (Combination therapy) | Baseline Up to Approximately Day 64
  The MTD and/or RP2D of ABBV-CLS-484 and VEGFR TKI will be determined during the combination therapy dose escalation phase of the study
Dose Expansion: Objective Response Rate (ORR) Of ABBV-CLS-484 Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Monotherapy) | Baseline Up to Approximately Day 42
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Dose Expansion: Objective Response Rate (ORR) Of ABBV-CLS-484 And PD-1 Targeting Agent Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Combination therapy) | Baseline Up to Approximately Day 64
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Dose Escalation: Objective Response Rate (ORR) Of ABBV-CLS-484 And VEGFR TKI Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Combination therapy) | Baseline Up to Approximately Day 64
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment

SECONDARY OUTCOMES:
Dose Escalation: Objective Response Rate (ORR) Of ABBV-CLS-484 Based On (RECIST) v1.1 (Monotherapy) | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Dose Escalation: Objective Response Rate (ORR) Of ABBV-CLS-484 And PD-1 Targeting Agent Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Combination therapy) | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment
Dose Escalation: Objective Response Rate (ORR) Of ABBV-CLS-484 And VEGFR TKI Based On Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 (Combination therapy) | Baseline through Study Completion (approximately 3 years)
  ORR is defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (30):
- United States (15):
  - University of Arizona Cancer Center - Tucson /ID# 262698, Tucson, Arizona
  - Yale University School of Medicine /ID# 225707, New Haven, Connecticut
  - Johns Hopkins Hospital /ID# 254056, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center /ID# 252009, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 249642, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 252010, Ann Arbor, Michigan
  - NYU Laura and Isaac Perlmutter Cancer Center - 34th Street /ID# 257869, New York, New York
  - Duke Cancer Center /ID# 251975, Durham, North Carolina
  - Carolina BioOncology Institute /ID# 225704, Huntersville, North Carolina
  - Perelman Center for Advanced Medicine /ID# 250188, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Ctr /ID# 225706, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 225705, Providence, Rhode Island
  - University of Texas Southwestern Medical Center /ID# 251974, Dallas, Texas
  - University of Texas MD Anderson Cancer Center /ID# 252004, Houston, Texas
  - NEXT Oncology /ID# 225708, San Antonio, Texas
- France (4):
  - Institut Paoli-Calmettes /ID# 260956, Marseille, Bouches-du-Rhone
  - IUCT Oncopole /ID# 252673, Toulouse, Occitanie
  - Centre Antoine-Lacassagne /ID# 252606, Nice, Provence-Alpes-Côte d'Azur Region
  - Hopital Foch /ID# 252607, Suresnes
- Israel (3):
  - Rabin Medical Center /ID# 263631, Petah Tikva, Central District
  - Hadassah Medical Center /ID# 252366, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 226756, Ramat Gan, Tel Aviv
- Japan (2):
  - National Cancer Center Hospital /ID# 225884, Chuo-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 252988, Wakayama, Wakayama
- South Korea (3):
  - Seoul National University Hospital /ID# 254635, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 260664, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 260665, Seoul
- Spain (3):
  - Institut Català d'Oncologia (ICO) - L'Hospitalet /ID# 252524, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 257374, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 228034, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baumgartner CK, Ebrahimi-Nik H, Iracheta-Vellve A, Hamel KM, Olander KE, Davis TGR, McGuire KA, Halvorsen GT, Avila OI, Patel CH, Kim SY, Kammula AV, Muscato AJ, Halliwill K, Geda P, Klinge KL, Xiong Z, Duggan R, Mu L, Yeary MD, Patti JC, Balon TM, Mathew R, Backus C, Kennedy DE, Chen A, Longenecker K, Klahn JT, Hrusch CL, Krishnan N, Hutchins CW, Dunning JP, Bulic M, Tiwari P, Colvin KJ, Chuong CL, Kohnle IC, Rees MG, Boghossian A, Ronan M, Roth JA, Wu MJ, Suermondt JSMT, Knudsen NH, Cheruiyot CK, Sen DR, Griffin GK, Golub TR, El-Bardeesy N, Decker JH, Yang Y, Guffroy M, Fossey S, Trusk P, Sun IM, Liu Y, Qiu W, Sun Q, Paddock MN, Farney EP, Matulenko MA, Beauregard C, Frost JM, Yates KB, Kym PR, Manguso RT. The PTPN2/PTPN1 inhibitor ABBV-CLS-484 unleashes potent anti-tumour immunity. Nature. 2023 Oct;622(7984):850-862. doi: 10.1038/s41586-023-06575-7. Epub 2023 Oct 4. PMID 37794185
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M20-431